CLINICAL TRIAL: NCT07119580
Title: Association Between Limbal Function and Tear Proteomics in Chronic Ocular Diseases: Focusing on Glaucoma
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Attending Physician, National Taiwan University Hospital
Other Study IDs: 202407137RINB
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma; Ocular Hypertension; Limbal Stem Cell Deficiency
Keywords: Corneal epithelium; Limbal stem cells; Glaucoma; Tear fluid; Proteome
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Limbal Stem Cell Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tear fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy control: Healthy control, without diagnosis of glaucoma.
- Glaucoma, newly diagnosed: Glaucoma patients who received topical antiglaucoma medications for less than 3 months.
- Glaucoma, long-term medication use: Glaucoma patients, received topical antiglaucoma medications for 1 year or longer.
- Glaucoma, unilateral: Patients with unilateral glaucoma or ocular hypertension and received treatment only in the diseased eye.

SUMMARY:
Background Intact corneal epithelium is important for the defense on the ocular surface, and the function of limbal stem cells is crucial to maintain its integrity. Certain chronic eye diseases, such as glaucoma, require long-term medication use. However, glaucoma patients often exhibit corneal punctate erosions and ocular surface inflammation. In cases where medication has been used for an extended period, patients may even show symptoms similar to limbal stem cell deficiency. Understanding how glaucoma medications affect the function of corneal limbal stem cells is a critical clinical issue.

Objectives To evaluate the effect of glaucoma and anti-glaucoma agents on corneal epithelial and limbal epithelial thickness as a surrogate of limbal stem cell function, and to understand the association between tear fluid proteome and limbal function in glaucoma patients.

Methods We planned to include 90 subjects with glaucoma, and analyze the absolute thickness and variation of corneal epithelium and limbal epithelium. Tear fluid samples will be collected and proteomic analysis will be performed to elucidate the association between protein.

Anticipated Results To elucidate the impact of different types and cumulative doses of glaucoma medications on the thickness of the corneal epithelium and limbal epithelium, and to understand the relationship between limbal function and tear proteomics in glaucoma patients. The expected results may help develop early detection methods for changes in corneal and limbal epithelial function and provide valuable insights for future research on drug design and the protection of limbal stem cells.

ELIGIBILITY:
Inclusion Criteria:

i. Age ≥ 18 years. ii. Healthy Control Group: No diagnosis of glaucoma or ocular hypertension. iii. Glaucoma, Newly Diagnosed Group: Diagnosed with angle-closure glaucoma, open-angle glaucoma, or ocular hypertension; antiglaucoma medication usage for less than 3 months.

iv. Glaucoma, Long-term Medication Group: Diagnosed with angle-closure glaucoma, open-angle glaucoma, or ocular hypertension; continuous use of intraocular pressure-lowering medications for more than 1 year.

v. Glaucoma, Unilateral Group: Diagnosed with unilateral glaucoma or ocular hypertension; only one eye receiving intraocular pressure-lowering treatment.

Exclusion Criteria:

i. History of severe ocular trauma, chemical burns, corneal ulcers, Stevens-Johnson syndrome with ocular involvement, or ocular graft-versus-host disease.

ii. History of corneal surgery, conjunctival surgery, trabeculectomy, or glaucoma drainage device implantation.

iii. Presence of ocular surface irregularity or limbal dysfunction due to conditions other than glaucoma or dry eye disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients in outpatient clinic setting.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Limbal epithelial thickness | Upon enrollment and at 6 months after enrollment (for newly diagnosed patients)
  Limbal epithelial thickness obtained from AS-OCT

SECONDARY OUTCOMES:
Corneal central epithelial thickness | Upon enrollment and at 6 months after enrollment (for newly diagnosed patients)
  Corneal epithelial thickness map obtained from AS-OCT
Proteomic findings of tear samples | Upon enrollment and at 6 months after enrollment (for newly diagnosed patients)
  Proteomic findings of tear samples

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsinchu Branch, Hsinchu, Taiwan